CLINICAL TRIAL: NCT00046722
Title: Effects of Marijuana on Neuropathic Pain in HIV-Related Peripheral Neuropathy: A Randomized, Double-Blind, Placebo-Controlled Study.
Brief Title: Marijuana for HIV-Related Peripheral Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Medicinal Cannabis Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C00-SF-101; CC# 056
Record Dates: First submitted 2002-10-01; First posted 2002-10-03 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Peripheral Nervous System Diseases; HIV Infections
Keywords: treatment experienced; complementary therapies; Neuropathy; Peripheral Neuropathy; HIV-Related Peripheral Neuropathy; HIV
MeSH Terms: conditions — Peripheral Nervous System Diseases; HIV Infections

INTERVENTIONS:
Drug: Smoked Marijuana

SUMMARY:
To evaluate whether smoked marijuana reduces pain in people with HIV-related peripheral neuropathy.

DETAILED DESCRIPTION:
The study will include subjects with peripheral neuropathy caused either by HIV-disease or antiretroviral medication for the treatment of HIV. A neurologist will conduct a neurological and pain evaluation to determine eligibility for the study. Subjects who meet all eligibility criteria will be admitted to the General Clinical Research Center at San Francisco General Hospital for seven days. Subjects will be randomized (like a toss of a coin) to smoke marijuana or a placebo (cigarettes with no THC).

ELIGIBILITY:
INCLUSION CRITERIA:

* HIV positive.
* Be 18 years or older.
* Diagnosis of HIV-related painful neuropathy.
* Stable antiretroviral therapy or no antiretroviral therapy for at least 8 weeks.
* Prior use of marijuana, at least 6 occasions in their lifetime prior to enrollment.

EXCLUSION CRITERIA: (Not allowed)

* Current use of smoked tobacco products.
* Current methadone treatment.
* Use of smoked marijuana within 30 days of enrollment.
* Diagnosis of diabetes mellitus.
* Currently receiving treatment with corticosteroids.
* Use of INH, dapsone or metronidazole within 8 weeks prior to enrollment.
* Severe heart disease, uncontrolled high blood pressure or lung disease.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Study Completion 2005-04

PRIMARY OUTCOMES:
Change in level of HIV-related neuropathic pain as recorded on a 100mm Visual Analog Scale.

SECONDARY OUTCOMES:
Change in level of experimentally-induced pain.

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Abrams, M.D., Principal Investigator — UCSF Community Consortium
Locations (1):
- University of California, San Francisco Community Consortium, San Francisco, California, United States

REFERENCES:
- [Result] Abrams DI, Jay CA, Shade SB, Vizoso H, Reda H, Press S, Kelly ME, Rowbotham MC, Petersen KL. Cannabis in painful HIV-associated sensory neuropathy: a randomized placebo-controlled trial. Neurology. 2007 Feb 13;68(7):515-21. doi: 10.1212/01.wnl.0000253187.66183.9c. PMID 17296917
- See also: Community Consortium — http://www.communityconsortium.org
- See also: Center for Medicinal Cannabis Research — http://cmcr.ucsd.edu